CLINICAL TRIAL: NCT04081961
Title: A Proof-of-concept, Open-label, Feasibility Study to Evaluate Mobile Applications and Biosensing (mHealth) Devices to Monitor Physical Activity and Respiratory Function in Smokers With and Without Respiratory Symptoms/COPD
Brief Title: Feasibility Study to Use Biosensing Devices to Monitor PA and Resp. Function in Smokers w and w/o Resp. Symptoms/COPD
Status: Completed | Type: Observational
Sponsor: Kazakhstan Academy of Preventive Medicine (Other)
Collaborators: Philip Morris International (Industry); Synergy Research Group (Industry)
Responsible Party: Sponsor
Other Study IDs: PMI.IIS.2016.1.
Record Dates: First submitted 2019-09-04; First posted 2019-09-09 (Actual); Results first posted 2020-01-09 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Signs and Symptoms, Respiratory; Mobile Applications; Activity Trackers; Respiratory Function Tests
MeSH Terms: conditions — Signs and Symptoms, Respiratory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Asymptomatic current smokers: No respiratory symptoms and preserved pulmonary function based on spirometry (FEV1/FVC of at least 0.70 after bronchodilation treatment and FVC ≥80% of the expected value)
  Interventions: Device: Anamed OEM device; Air Next mobile spirometry device
- "Grey zone" current smokers: Initially preserved pulmonary function based on spirometry, but with clinical symptoms based on COPD Assessment Test (CAT≥10) and results of the 6-min walk test (6 MWT) less than 450 meters.
  Interventions: Device: Anamed OEM device; Air Next mobile spirometry device
- Current smokers with COPD: Current smokers with a confirmed diagnosis of COPD (GOLD stage I-III)
  Interventions: Device: Anamed OEM device; Air Next mobile spirometry device

INTERVENTIONS:
Device: Anamed OEM device; Air Next mobile spirometry device — Anamed OEM (Original Equipment Manufacturer) device - physical activity and vital signs monitoring; Air Next mobile spirometry device

SUMMARY:
This study examines the feasibility and acceptability of using mobile applications and biosensing (mHealth) devices in detecting vitality parameters in current smokers with and without respiratory symptoms/COPD (e.g., heart rate, blood oxygenation, steps/motion) for a future big-scale study.

DETAILED DESCRIPTION:
The study is designed to investigate feasibility of using mHealth devices to improve the treatment, assessment, compliance, and outcomes in smokers with and without respiratory symptoms/COPD. The study aims to reveal and address the anticipated barriers to the acceptance and implementation of mHealth devices in this patient population and clinical setting. As is well documented, the more attention patients receive from medical personnel, the better their clinical outcomes. Here we are attempting to use device-driven monitoring applications, interactive reminders, and teaching modules to deliver a constant positive feedback loop to patients to improve their health decisions.

Objectives of the study:

To assess the feasibility of using mHealth devices in current smokers with and without respiratory symptoms/COPD.

To assess the utility (i.e., validity and reproducibility) of mHealth devices in detecting vitality parameters in current smokers with and without respiratory symptoms/COPD (e.g., heart rate; blood oxygenation; steps/motion; FEV1, FVC, and their ratio; peak expiratory flow [PEF]).

ELIGIBILITY:
Inclusion Criteria:

* Current smokers who are currently smoking conventional cigarettes with a minimum of 10 pack-year smoking history
* Able to use and willing to be trained to use mHealth devices

Exclusion Criteria:

* COPD exacerbation that has not resolved at least 28 days prior to screening
* COPD exacerbation occurring after screening but before the first study visit
* Pneumonia or other respiratory tract infections that have not resolved at least 14 days prior to screening
* Pneumonia occurring after screening but before the first study visit
* Active respiratory disorders: tuberculosis, lung cancer, significant bronchiectasis, sarcoidosis, bronchial asthma, lung fibrosis, pulmonary hypertension, interstitial lung diseases, or other active pulmonary diseases
* Any co-morbid medical condition that in the opinion of the investigator would make participation in the study unsafe or unfeasible, including conditions that prohibit completion of exercise testing
* Use of supplemental oxygen therapy
* Inability to abstain from smoking during the period in which the participant is admitted to the Kazakhstan Academy of Preventive Medicine (KAPM) COPD Center
* A history of allergy or hypersensitivity to metal, particularly stainless steel
* Any vital sign indicator, for example, hypertension or tachycardia at rest that, at the discretion of the investigator, would make participation in the study unsafe or unfeasible
* Women who test positive for pregnancy during screening, lactating women, or women planning on becoming pregnant during the study
* Participants using assistive devices like walking aids, as these are likely to interfere with physical activity

Ages: 40 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Residents of City of Almaty aged 40-59 who smoke conventional cigarettes with a minimum of 10 pack-year smoking history
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2019-06-07 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Almaz Sharman, Dr, Principal Investigator — Kazakhstan Academy of Preventive Medicine
Locations (1):
- Kazakhstan Academy of Preventive Medicine, Almaty, Kazakhstan

IPD SHARING:
Plan to Share IPD: Yes
The dataset after the re-identification will be available to other researchers on the 'www.intervals.science' platform.
Supporting Information: Study Protocol
Time Frame: Data will be available after May 1, 2020 without time limit.
URL: http://www.intervals.science

REFERENCES:
- [Derived] Sharman A, Zhussupov B, Sharman D, Kim I. Evaluating Mobile Apps and Biosensing Devices to Monitor Physical Activity and Respiratory Function in Smokers With and Without Respiratory Symptoms or Chronic Obstructive Pulmonary Disease: Protocol for a Proof-of-Concept, Open-Label, Feasibility Study. JMIR Res Protoc. 2020 Mar 26;9(3):e16461. doi: 10.2196/16461. PMID 32213479

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Asymptomatic Current Smokers | "Grey Zone" Current Smokers | Current Smokers With COPD
Started | 9 | 9 | 9
Completed | 9 | 9 | 9
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Asymptomatic Current Smokers | "Grey Zone" Current Smokers | Current Smokers With COPD | Total
Number analyzed (Participants) | 9 | 9 | 9 | 27
Age, Continuous [Mean (Full Range); unit: years] | 50.9 [44 to 58] | 50.8 [42 to 58] | 51.4 [44 to 59] | 51.0 [42 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 6
  Male | 7 | 7 | 7 | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Kazakhstan | 9 | 9 | 9 | 27

OUTCOME MEASURES:

1. Primary Outcome: Rate of Recruitment
Description: Recruitment is defined as the number of potential participants screened for study eligibility versus the number of persons who enrolled in the study.
Time Frame: Baseline
Population: The number of potential participants screened for study eligibility
Measure: Count of Participants; unit: Participants
Arm/Group | Asymptomatic Current Smokers | "Grey Zone" Current Smokers | Current Smokers With COPD
Number analyzed (Participants) | 29 | 27 | 21
Participants | 9 | 9 | 9

2. Primary Outcome: Rate of Retention
Description: Retention is defined as the proportion of participants enrolled who completed the intervention and all study measures.
Time Frame: through study completion, an average of 90 days
Population: Participants recruited to the study
Measure: Count of Participants; unit: Participants
Arm/Group | Asymptomatic Current Smokers | "Grey Zone" Current Smokers | Current Smokers With COPD
Number analyzed (Participants) | 9 | 9 | 9
Participants | 9 | 9 | 9

3. Primary Outcome: Protocol Adherence
Description: Adherence to the study protocol is determined as the proportion of participants enrolled from whom all mHealth parameters registered every day.
Time Frame: through study completion, an average of 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Asymptomatic Current Smokers | "Grey Zone" Current Smokers | Current Smokers With COPD
Number analyzed (Participants) | 9 | 9 | 9
Participants | 4 | 5 | 8

ADVERSE EVENTS:
Time Frame: 90 days after participant was recruited to the study
Arm/Group | Asymptomatic Current Smokers | "Grey Zone" Current Smokers | Current Smokers With COPD
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-06-03): https://cdn.clinicaltrials.gov/large-docs/61/NCT04081961/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-14): https://cdn.clinicaltrials.gov/large-docs/61/NCT04081961/SAP_001.pdf